CLINICAL TRIAL: NCT01851044
Title: The Treatment of Lateral Epicondylitis: the Effect of Platelet Rich Plasma on Healing -- A Randomized Controlled Double-Blinded Trial
Brief Title: The Effect of Platelet Rich Plasma on Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Hatanpää City Hospital, Tampere, Finland (Unknown)
Responsible Party: Principal Investigator, Olli Leppänen, Researcher, Tampere University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R11031
Record Dates: First submitted 2013-05-05; First posted 2013-05-10 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Lateral Epicondylitis; Elbow Pain
Keywords: Platelet Rich Plasma; Whole Blood Injection; Lateral Epicondylitis; Tennis Elbow
MeSH Terms: conditions — Tennis Elbow | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vehicle (Saline) (Placebo Comparator): 2 ml of saline is injected to the proximal insertion of extensor carpi radialis brevis (ECRB) muscle.
  Interventions: Procedure: Platelet Rich Plasma
- Whole Blood (Active Comparator): 2 ml of patient own venous blood is injected to the proximal insertion of ECRB.
  Interventions: Procedure: Whole Blood Injection
- Platelet Rich Plasma (Experimental): 9 ml of patient own venous blood is centrifuged using The Arthrex ACP® Double Syringe System and 2 ml of platelet rich plasma is injected to the proximal insertion of ECRB.
  Interventions: Procedure: Saline Injection

INTERVENTIONS:
Procedure: Platelet Rich Plasma
  Arms: Vehicle (Saline)
Procedure: Whole Blood Injection
  Arms: Whole Blood
Procedure: Saline Injection
  Arms: Platelet Rich Plasma

SUMMARY:
The purpose of this study is to compare the effects of platelet rich plasma, whole blood and saline vehicle on the natural course of lateral epicondylitis.

DETAILED DESCRIPTION:
Lateral epicondylitis, also known as "tennis elbow", is the most common work-related disease of the upper extremity. Usually it has favorable natural healing-tendency, but sometimes it is responsible for long-lasting disability. The pathogenesis of this disease has remained unclear, however it has been speculated that the role of inflammation is smaller than previously believed. Instead, anatomical and vascular factors may play a much greater role. The evidence for the operative treatment is lacking, and the conservative treatment is therefore preferred. The conservative treatment used to rely largely on corticosteroid injections to the extensor muscle insertions. However, it has been shown that corticosteroids, in fact, tend to increase the subjective pain in the long run. Several studies -- most of them unfortunately underpowered -- have been carried out to find an efficient conservative treatment to this disease, but none of them has turned out to be significantly better than others. During the last couple of years, platelet rich plasma (PRP) has been used as a treatment in several musculoskeletal diseases (e.g. fracture healing, cartilage regeneration, wound healing). PRP is a substance centrifuged from patient own blood. There are a couple of studies regarding the use of PRP in lateral epicondylitis. The results are mostly positive; however it has not been thoroughly shown that it would be more effective than patient's whole blood. The hypothesis of this study is that PRP is more effective in the treatment of lateral epicondylitis than whole blood or saline vehicle injection. The primary outcome measures are pain (VAS) and the Disabilities of the Arm, Shoulder and Hand -score (DASH).

ELIGIBILITY:
Inclusion Criteria:

* The duration of symptoms over 3 months
* Primary conservative treatment (physiotherapy, NSAID, ...) has been tried

Exclusion Criteria:

* Significant systemic diseases
* Any surgical operation of the particular elbow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-02; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Pain (Visual Analog Scale) | 52 weeks

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand -score | 52 weeks

OTHER OUTCOMES:
Grip strength (Jamar) | 52 weeks
Need for non-steroidal anti-inflammatory drugs (NSAID) | 52 weeks
The duration of the potential sick leave due to lateral epicondylitis | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hatanpää City Hospital, Tampere, Finland

REFERENCES:
- [Derived] Karjalainen TV, Silagy M, O'Bryan E, Johnston RV, Cyril S, Buchbinder R. Autologous blood and platelet-rich plasma injection therapy for lateral elbow pain. Cochrane Database Syst Rev. 2021 Sep 30;9(9):CD010951. doi: 10.1002/14651858.CD010951.pub2. PMID 34590307